CLINICAL TRIAL: NCT01204047
Title: Wheelchair Propulsion Function and Physical Capacity in Persons With Spinal Cord Injury
Brief Title: Wheelchair Mobility Assessment of Individuals With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Other Study IDs: TMP-MN-007
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The specific aims of this study are: 1) to assess the test-retest reliability of a modification of an existing wheelchair propulsion assessment and 2) validate the modification against traditional measures of physical strength, power, and endurance in a group of persons with spinal cord injury (SCI).

DETAILED DESCRIPTION:
The ability to independently self-propel and transfer oneself is a crucial component of daily life for individuals with a spinal cord injury. This ability is related in part to an individual's strength, power, and endurance, but it is unknown which of these measures is most important to achieve a high level of wheelchair function. Identification of which physical performance parameters are best related to wheeled mobility performance is essential in developing interventions to improve said performance. Currently, clinic-friendly assessments of a person's wheeled mobility ability do not exist. We have developed a modified, clinic-friendly version of validated wheelchair mobility assessment that can be completed in most clinics. Before it can be implemented by clinicians its reliability must be established. Crossvalidating it against standard measures of physical performance will allow for the identification of the most appropriate exercise interventions to improve independent wheeled mobility.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury
* American Spinal Injury Association Impairment Scale (AIS) A-D
* Self-reported ability to self-propel themselves in a manual wheelchair
* Age 18 or older

Exclusion Criteria:

* surgery within 6 months
* pressure ulcer within 3 months
* upper limb pain that limits completion of exercise
* recurrent acute infection or illness requiring hospitalization or IV antibiotics
* pregnancy
* previous myocardial infarction or cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2008-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Ability Score | within a 14 day period
  The ability score is the sum of the number of items successfully completed in the wheelchair propulsion assessment. There are 8 items in the assessement, which will be completed in the following order: 1) Figure of 8 Shape, 2) Doorstep Crossing, 3) Platform Ascent, 4) 15 meter sprint, 5) Ramp Ascent (5% grade), 6) Ramp Ascent (8% grade), 7) 150 meter propulsion, and 8) Timed Level Transfer.

SECONDARY OUTCOMES:
Muscular strength | 1 day
  Upper extremity dynamic strength testing will be performed on a Helms equalizer 1000 multi-station exerciser using the following maneuvers: overhead press, horizontal row, vertical butterfly, biceps curl, latissimus pull down (either to the chest or neck), and dips. The 1-repetition maximum (1-RM) will be calculated using the Mayhew regression equation.
Anaerobic power | 1 day
  Participants will propel a table-mounted Monark 894e ergometer for 30 seconds at maximal speed against constant force. The constant resistance for each subject will be set at 1.5% and 3.5% of their body mass, for tetraplegia and paraplegia respectively. Data for three variables will be obtained: a) peak power, defined as the highest average mechanical power measured during any 5-second period, b) mean power, the average power sustained during the 30-second test period, and c) rate of fatigue, defined as the degree of power drop-off during the test.
Cardiovascular endurance | 1 day
  Endurance will be measured using a calibrated upper arm ergometer. An initial exercise workload of 0 Watts at 60 revolutions per minute (RPM) for three minutes will be followed by three minute stages increasing in 20 Watt increments. Responses to exercise will be continuously monitored via open-circuit spirometry and 12-lead electrocardiography. Peak Work will be defined as volitional fatigue, inability to maintain targeted workload, or the point at which increasing workload fails to further increase VO2.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami Miller School of Medicine, The Miami Project to Cure Paralysis
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States